CLINICAL TRIAL: NCT05110586
Title: The Effect of Different Electrical Stimulations on Pain, Functional Capacity and Quality of Life in Multiple Sclerosis Patients
Brief Title: Electrical Stimulations on Pain, Functional Capacity and Quality of Life in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, Asst. Prof., Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ipekkirmaci
Record Dates: First submitted 2021-10-14; First posted 2021-11-08 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
Keywords: pain; functional capacity; Quality of life; electrotherapy
MeSH Terms: conditions — Multiple Sclerosis; Pain | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st group: TENS (Experimental): Tens will be applied.
  Interventions: Other: Electrotherapy
- 2nd group: Interferential current (Experimental): Interferential current will be applied.
  Interventions: Other: Electrotherapy

INTERVENTIONS:
Other: Electrotherapy — Applications will be applied for 4 weeks, 5 days a week

SUMMARY:
Multiple Sclerosis (MS) is a chronic neurological disease with local inflammation, gliosis and demyelination in the central nervous system (CNS). It is characterized by demyelinating plaques in the brain and spinal cord. Many different symptoms can be seen in the CNS, depending on the affected areas. One of the most common symptoms in these patients is pain. Approximately 50% of patients complain of pain at some point in their lives, and pain is one of the initial symptoms in 20%. Pain may originate from the musculoskeletal system; It may also develop due to inflammation and upper motor neuron damage and may have a neuropathic character . In conclusion, pain in MS negatively affects the physical and emotional functions and quality of life of patients.

In addition to pharmacological treatments, non-pharmacological interventions such as electrotherapy and exercise are present among the available treatments for pain in MS patients.

DETAILED DESCRIPTION:
In electrotherapy applications, Transcutaneous Electrical Nerve Stimulation (TENS) is defined as a method of applying high-frequency low-intensity electric current to the nervous system through superficial electrodes placed on the painful area or the nerve innervating that area, used all over the world in the treatment of pain, FDA approved in the United States.

Its effectiveness is thought to be the result of a combination of effects such as stimulation of large-scale afferent fibers that inhibit the activity of primary afferent pain neurons or endogenous opioid-dependent mechanisms including the release of dynorphins, enkephalins and endorphins in the central nervous system .

Interferential current are medium frequency currents. The analgesic effect of this current is based on the gate control theory. The disadvantage compared to TENS is that it provides lower neural adaptations with higher currents.

As a result of this study, it is thought that the determination of effective treatment methods for pain, which is one of the common symptoms of MS patients, will increase the functional capacity and quality of life of the patient.

In the study, patients who meet the inclusion criteria will be divided into 2 groups by randomization, TENS will be applied to the 1st group, and interference current will be applied to the 2nd group. Applications will be applied for 4 weeks, 5 days a week. Evaluations will be made by a blind physiotherapist twice, before and after the treatment. Assessments include sociodemographic information, pain, functional capacity, and quality of life.

In addition to the studies in the literature, this study will be the first to compare the effectiveness of different electrical stimulations in pain in MS.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with MS according to McDonald 2010 diagnostic criteria
* 18-65 years old
* Volunteering to participate in the study

Exclusion Criteria:

* Less than 18 years old, over 65 years old
* Having a history of trauma in the last 1 year
* Having alcohol and substance addiction
* Having diabetes mellitus
* Presence of other known neurological disease
* Having a pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) | Change from Baseline at 4 weeks
  The Visual Analog Scale (VAS) is a scale used to determine the severity of pain. Two end definitions of the parameter to be evaluated are written on the two end points of a 100 mm line and the patient is asked to indicate where his/her condition is appropriate on this line.
Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain questionnaire | Change from Baseline at 4 weeks
  The scale is scored between 0-24 points and above 12 points suggests neuropathic pain.

SECONDARY OUTCOMES:
2 min walk test | Change from Baseline at 4 weeks
  Individuals are asked to walk as fast as possible in a 25 m corridor without running. The distance they walked for two minutes is recorded.
Multiple Sclerosis International Quality of Life Questionnaire | Change from Baseline at 4 weeks
  The questionnaire indicates quality of life. the index score are linearly transformed and standardized on a 0 to 100 scale, where 0 indicates the worst possible level of QoL and 100 indicates the best level.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katirci Kirmaci ZI, Adiguzel H, Gogremis M, Kirmaci YS, Inanc Y, Tuncel Berktas D. The effect of Transcutaneous Electrical Nerve Stimulation (TENS) and Interferential Currents (IFC) on pain, functional capacity, and quality of life in patients with multiple sclerosis: A randomized controlled, single-blinded study. Mult Scler Relat Disord. 2023 Mar;71:104541. doi: 10.1016/j.msard.2023.104541. Epub 2023 Jan 29. PMID 36738692